CLINICAL TRIAL: NCT01125488
Title: Maintenance Therapy of LNG-IUS in Conjunction With the GnRH Agonist to Prevent the Recurrence of Symptomatic Endometriosis After Conservative Surgery: A Prospective Randomized, Phase III Trial
Brief Title: Maintenance Therapy of Levonorgestrel-releasing Intrauterine System (LNG-IUS) to Prevent the Recurrence of Symptomatic Endometriosis After Conservative Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Yi-Jen Chen MD, Department of Obstetrics & Gynecology,Taipei Veterans General Hospital,Taiwan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VGHIRB 97-04-03
Record Dates: First submitted 2010-04-26; First posted 2010-05-18 (Estimated); Last update posted 2010-06-08 (Estimated); Status verified 2010-06

CONDITIONS: Endometriosis
Keywords: Maintenance therapy; LNG-IUS; recurrence,endometriosis; Recurrence
MeSH Terms: conditions — Endometriosis; Recurrence | interventions — Gonadotropin-Releasing Hormone; Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LNG-IUS (Experimental): LNG-IUS insertion during conservative surgery and GnRH agonist 6 doses.
  Interventions: Device: LNG-IUS; Drug: GnRH agonist (triptorelin)
- GnRH agonist (Active Comparator): The second group of patients receive GnRH agonist (triptorelin 3.75 mg, sc q28day) alone for 24 weeks.
  Interventions: Drug: GnRH agonist (triptorelin)

INTERVENTIONS:
Device: LNG-IUS — levonorgestrel-releasing intrauterine system (LNG-IUS) 52mg, duration 5 years
  Other Names: mirena
  Arms: LNG-IUS
Drug: GnRH agonist (triptorelin) — GnRH agonist (triptorelin 3.75 mg, sc q28day)

SUMMARY:
The recurrence rates of endometriosis reported in women 5 years after therapy with gonadotropin releasing hormone (GnRH) agonist were 74% for severe disease . No strategies to prevent the recurrence of endometriosis have been uniformly successful. Local progesterone treatment of endometriosis-associated dysmenorrhea with a levonorgestrel-releasing intrauterine system (LNG-IUS) for 12 months has resulted in a significant reduction in dysmenorrhea, pelvic pain and dyspareunia; a high degree of patient satisfaction; and a significant reduction in the volume of rectovaginal endometriotic nodules. LNG-IUS may become a more important option if a long-term medical suppression of endometriosis.

Based on literature review, I hypothesized that maintenance therapy of LNG-IUS in conjunction with the GnRH agonist could lower the recurrence rates endometriosis after conservative surgery. We try to answer the question whether maintenance therapy of LNG-IUS in conjunction with the GnRH agonist could lower the recurrence rates and thus extend the symptom-free interval (menorrhagia and dysmenorrhea) as compared to GnRH agonist alone after conservative surgery in severe endometriosis cases.

DETAILED DESCRIPTION:
Participants:

This post-surgical medical therapy trial will be undertaken among patients with moderate-severe symptomatic endometriosis (rASRM score >16, according to the American Society for Reproductive Medicine) or adenomyosis. Symptomatic endometriosis means menorrhagia or dysmenorrhea. All patients were surgically treated by a conservative approach (means preserve uterus and ovary).

Interventions:

In all patients, were prescribed 600 mg elemental Ca and 400 IU vitamin D (bid). The first group of patients receive LNG-IUS for 5 years and GnRH agonist (triptorelin 3.75 mg, sc q28day) for 24 weeks.

The second group of patients receive GnRH agonist (triptorelin 3.75 mg, sc q28day) alone for 24 weeks.

Patients were evaluated every month for 24 weeks, and at 3,6,9,12,15,18,21,24 months after the end of medical treatment.

Objectives and outcomes:

The main objective of this trial was to assess the clinical efficacy of LNG-IUS maintenance therapy to prevent recurrence of endometriosis. Thus the primary outcome measures of this trial is the recurrence rate of endometriosis.

During this trial, recurrence was defined as elevation of CA125 (6) or endometriosis lesion in sonography or symptoms suggesting endometriosis including menorrhagia or dysmenorrhea.

The pain score diary was based on the visual analogue scale in which patients recorded the occurrence an intensity of their pain daily. VAS consists of a subjective evaluation of the pain on a scale of 10 in which 0 is no pain and 10 the most severe pain (7).

Bleeding and menorrhagia were assessed as: 0= no bleeding; 1=spotting (light bleeding not requiring sanitary protection); 2=light bleeding (light bleeding requiring sanitary protection); 3=normal bleeding (bleeding similar to normal menstrual blood flow); and 4=heavy bleeding (bleeding exceeding normal menstrual blood flow). No bleeding was defined as 30 consecutive days with bleeding score 0 (8).

Randomization process:

Treatment allocation was performed in accordance with a computer-generated randomization sequence using numbered, sealed envelopes.

Evaluation of efficacy:

Sample size:

In calculating the sample size required, the primary assessment was the recurrence rates. A 31% recurrence rate after laparoscopic reproductive surgery and post-surgical treatment with a GnRH agonist has been reported (9). We expected a decrease in recurrence rates after laparoscopic conservative surgery and post-surgical treatment with GnRH agonist plus LNG-IUS. A difference of 25% between the allocated treatments was considered significant. To have a 90% chance of detecting such a difference at an overall significant level of 5%, 40 patients for each group were required.

Endpoints:

We will follow the patients for 2 years, after the end of GnRH agonist medical treatment. Thus the primary outcome measures of this trial is the recurrence rate of endometriosis.

The main objective of this trial was to assess the clinical efficacy of LNG-IUS maintenance therapy to prevent recurrence of endometriosis.

Statistical analysis plan:

The cumulative proportion of recurrences by plotting percent recurrences as a function of time was estimated by the method of Kaplan and Meier. The survival curves for each allocated treatment were compared with the log-rank test.

For quantitative variables with normal distribution, the parametric t-test was used; in the case of the other variables, the non-parametric Mann-Whitney test was applied. For qualitative variables, x2-test or Fisher's exact test were used. For dependent variables with numerical scores referring to long-term measurement, multivariate analysis of variance ( MANOVA) was used.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate-severe symptomatic endometriosis (rASRM score >16) according to the American Society for Reproductive Medicine) or adenomyosis. Symptomatic endometriosis means menorrhagia or dysmenorrhea.
* All patients were surgically treated by a conservative approach.
* Levels of serum CA125 is higher than normal range.

Exclusion Criteria:

* Further desire for child bearing in future 3 years.
* Any treatment for endometriosis within the previous 2 months.
* Any concomitant disease that can be an established cause of chronic pelvic pain and anemia (Thalassemia anemia, inflammation sequela, myoma , and pelvic congestion etc)

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-03 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of endometriosis | 2 years
  We will follow the patients for 2 years, after the end of GnRH agonist medical treatment. Number of Participants with recurrence as a Measure of the clinical efficacy of LNG-IUS maintenance therapy to prevent recurrence of endometriosis.

SECONDARY OUTCOMES:
the safety of LNG-IUS maintenance therapy to prevent recurrence of endometriosis. | 2 years
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Jen Chen, MD, Principal Investigator — Department OBS & GYN, Taipei Veterans General Hospital
Locations (1):
- Taipei Veterans Genreal Hospital, Taipei, Taiwan